CLINICAL TRIAL: NCT01668355
Title: PACT to Improve Health Care in People With Serious Mental Illness (SMI-PACT)
Brief Title: PACT for Individuals With Serious Mental Illness
Acronym: SMI-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDP 12-177
Record Dates: First submitted 2012-08-07; First posted 2012-08-20 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia Spectrum & Other Psychotic Disorders
Keywords: Delivery of Healthcare; Health Services Research; Integrated Healthcare Systems; Healthcare Quality, Access, and Evaluation; Primary Care; Quality Improvement; Psychotic Disorders; Medical Home; Psychiatry; Patient Care Management; Nursing Care Management; Treatment Costs
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: medical home tailored for people with serious mental illness
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMI-PACT (Experimental): Patient Aligned Care Team (PACT) medical home model to address the physical healthcare needs of individuals with serious mental illness
  Interventions: Other: Patient Aligned Care Team (PACT)
- Usual Care (No Intervention): Usual Primary Care

INTERVENTIONS:
Other: Patient Aligned Care Team (PACT) — An integrated healthcare model to coordinate and address physical health needs of people with serious mental illness. This specialized PACT medical home model is designed for individuals with serious mental illness.
  Other Names: SMI-PACT
  Arms: SMI-PACT

SUMMARY:
People with serious mental illness have difficulty making good use of primary care, and die, on average, years earlier than others in the population. The greatest contributors to this premature mortality are medical illnesses, especially cardiovascular disease and cancer. The Patient Centered Medical Home is a model for reorganizing primary care practice so that healthcare is more effective, efficient, and user-friendly. It has been implemented across VA as the, "Patient Aligned Care Team" (PACT). It is unclear, however, how this PACT model applies to people whose predominant illness is treated by specialists. This is the case for people with serious mental illness (SMI), many of whom receive ongoing treatment at mental health clinics. To achieve optimal health outcomes in the population with SMI, it may be necessary to adapt the PACT model so that it includes approaches that have proven to improve healthcare in this population. This project implements an adapted "SMI-PACT" model, and evaluates its effect on Veterans with SMI.

DETAILED DESCRIPTION:
Background/Rationale:

People with serious mental illness (SMI) die, on average, many years prematurely, with rates of premature mortality 2 to 3 times greater than the general population. Over 60% of premature deaths in this population are due to "natural causes," especially poorly treated cardiovascular, respiratory, and infectious diseases. Although the VA is a centrally organized, comprehensive healthcare system, Veterans with SMI still have difficulty navigating the system, and are at substantially elevated risk for premature death. Too often, they do not attend scheduled appointments or fail to engage in primary care treatment, and consequently do not get valuable preventive and primary care services.

Primary care in VA has undergone significant transformation under the Patent Aligned Care Team (PACT) model, which is based on the Patient Centered Medical Home (PCMH) concept. PACT has the goal of improving the quality, efficiency, and patient-centeredness of primary care. But it remains unclear how PACT will impact the large populations of Veterans whose predominant illness is treated in specialty settings, such as people with SMI. Research can inform efforts to apply the PACT model. For example, while people with SMI do poorly with usual primary care arrangements, there is substantial evidence that integrated care and medical care management approaches can improve medical treatment and outcomes, and reduce treatment costs, in people with SMI.

Objective:

Using available evidence, the investigators propose to implement and evaluate a specialized PACT model that meets the needs of individuals with SMI ("SMI-PACT").

Methods:

This project will partner with leadership to implement SMI-PACT, with the goal of improving healthcare and outcomes among people with SMI, while reducing unnecessary use of emergency and hospital services. Evidence-based quality improvement strategies will be used to reorganize processes of care. In a site-level controlled trial, this project will evaluate the effect, relative to usual care, of SMI-PACT implementation on (a) provision of appropriate preventive and medical treatments; (b) patient health-related quality of life and satisfaction with care; and (c) medical and mental health treatment utilization and costs. The project includes a mixed methods formative evaluation of usual care and SMI-PACT implementation to strengthen the intervention, and assess barriers and facilitators to its implementation. Mixed methods will also be used to investigate the relationships between organizational context, intervention factors, and patient and provider outcomes; and identify patient factors related to successful patient outcomes.

Significance:

This project's approach to SMI-PACT is consistent with the VA PACT model, and with efforts in VA to improve care for Veterans with psychiatric disorders. This will be one of the first projects to systematically implement and evaluate the PCMH and PACT concepts for patients with serious mental illness. Should SMI-PACT be demonstrated to be feasible and effective, the model could be used more broadly to improve the quality and efficiency of care for Veterans.

ELIGIBILITY:
Inclusion Criteria:

Patient subjects:

* currently enrolled at one of the 3 participating VA healthcare centers
* Veteran
* diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, chronic severe PTSD, or recurrent major depression with psychosis
* Milestone of Recovery Scale (MORS) score is 6 or above (indicates recovery status is coping rehabilitating or better)

Staff subjects:

* employed at one of the 3 participating VA healthcare centers
* member of PACT, member of SMI PACT, member of primary care mental health integration, provider at mental health clinic, administrator overseeing mental health, or administrator overseeing primary care

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Young, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (3):
- United States (3):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Young AS, Cohen AN, Chang ET, Flynn AWP, Hamilton AB, Oberman R, Vinzon M. A clustered controlled trial of the implementation and effectiveness of a medical home to improve health care of people with serious mental illness: study protocol. BMC Health Serv Res. 2018 Jun 7;18(1):428. doi: 10.1186/s12913-018-3237-0. PMID 29880047
- [Derived] Young AS, Chang ET, Cohen AN, Oberman R, Chang DT, Hamilton AB, Lindamer LA, Sanford J, Whelan F. The Effectiveness of a Specialized Primary Care Medical Home for Patients with Serious Mental Illness. J Gen Intern Med. 2022 Oct;37(13):3258-3265. doi: 10.1007/s11606-021-07270-x. Epub 2022 Apr 5. PMID 35380346

RESULTS

PARTICIPANT FLOW:
Groups:
- SMI-PACT: Patient Aligned Care Team (PACT) medical home to address the physical healthcare needs for individuals with serious mental illness (SMI).
  An integrated healthcare model designed to coordinate and address physical health needs of people with serious mental illness.
Period: Overall Study
Arm/Group | SMI-PACT | Usual Care
Started | 164 | 167
Completed | 155 | 165
Not Completed | 9 | 2
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- SMI-PACT: Patient Aligned Care Team (PACT) medical home model to address the physical healthcare needs for individuals with serious mental illness (SMI). An integrated healthcare model to coordinate and address physical health needs.
- Total: Total of all reporting groups
Arm/Group | SMI-PACT | Usual Care | Total
Number analyzed (Participants) | 164 | 167 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.4) | 54.5 (13.9) | 56.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 31 | 45
  Male | 150 | 136 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 19 | 41
  Not Hispanic or Latino | 138 | 127 | 265
  Unknown or Not Reported | 4 | 21 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 74 | 37 | 111
  White | 59 | 94 | 153
  More than one race | 8 | 11 | 19
  Unknown or Not Reported | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Provision of Appropriate Preventive and Medical Treatments
Description: Screened for body mass index, blood pressure, lipids, and glucose or hemoglobin A1c.
Time Frame: 15 months
Population: These are the number of subjects for whom data was available for this measure during the relevant time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | SMI-PACT | Usual Care
Number analyzed (Participants) | 164 | 166
Participants
  Screened for Body Mass Index | 144 | 117
  Screened for Blood Pressure | 146 | 131
  Screened for Lipids | 88 | 41
  Screened for Glucose or Hemoglobin A1c | 119 | 85

2. Primary Outcome: Patient Health-related Quality of Life: Veterans RAND 6 Item Health Survey (VR-6) Physical Health
Description: Physical health related quality of life. The scale range is 0 to 100. Higher scores mean a better outcome.
Time Frame: 15 months
Population: These are the number of subjects for whom data was available for this measure during the relevant time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMI-PACT | Usual Care
Number analyzed (Participants) | 129 | 133
score on a scale | 38.9 (11.0) | 37.2 (11.6)

3. Primary Outcome: Patient Health-related Quality of Life: Veterans RAND 6 Item Health Survey (VR-6) Mental Health
Description: Mental health related quality of life. The scale range is 0 to 100. Higher scores mean a better outcome.
Time Frame: 15 months
Population: These are the number of subjects for whom data was available for this measure during the relevant time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMI-PACT | Usual Care
Number analyzed (Participants) | 129 | 133
score on a scale | 42.3 (12.3) | 37.6 (12.8)

4. Primary Outcome: Patient Satisfaction With Care: Ambulatory Care Experiences Survey (ACES; Short Form)
Description: Evaluates patients' experiences and satisfaction with a physician's practice. The ACES uses the Institute of Medicine definition of primary care as its underlying conceptual model for measurement. The ACES range is 0 to 100. Higher scores mean a better outcome.
Time Frame: 15 months
Population: These are the number of subjects for whom data was available for this measure during the relevant time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMI-PACT | Usual Care
Number analyzed (Participants) | 152 | 155
score on a scale | 68 (24.2) | 66.7 (25.1)

5. Primary Outcome: Patient Satisfaction With Care: Patient Assessment of Chronic Illness Care (ACIC/PACIC)
Description: Assesses the patient's experience and satisfaction with receipt of chronic care. This measure aligns with the Chronic Care Model. The ACIC/PACIC ranges from from 1 to 5. Higher scores mean a better outcome.
Time Frame: 15 months
Population: These are the number of subjects for whom data was available for this measure during the relevant time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMI-PACT | Usual Care
Number analyzed (Participants) | 134 | 130
score on a scale | 2.7 (1.0) | 2.9 (1.0)

6. Other Pre Specified Outcome: Patient Psychopathology: Behavior and Symptom Identification Scale (BASIS-R) Psychosis
Description: Assesses patient psychopathology in the domain of psychosis. Scores range from 0 to 4. Higher scores mean a worse outcome.
Time Frame: 15 months
Population: These are the number of subjects for whom data was available for this measure during the relevant time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMI-PACT | Usual Care
Number analyzed (Participants) | 164 | 165
score on a scale | 0.88 (0.79) | 0.65 (0.71)

7. Other Pre Specified Outcome: Patient Psychopathology: Behavior and Symptom Identification Scale (BASIS-R) Depression Daily Functioning
Description: Assesses patient psychopathology in the domain of depression/daily functioning. Scores range from 0 to 4. Higher scores mean a worse outcome.
Time Frame: 15 months
Population: These are the number of subjects for whom data was available for this measure during the relevant time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMI-PACT | Usual Care
Number analyzed (Participants) | 164 | 165
score on a scale | 1.63 (0.68) | 1.71 (0.72)

8. Other Pre Specified Outcome: Patient Psychopathology: Behavior and Symptom Identification Scale (BASIS-R) Interpersonal Functioning
Description: Assesses patient psychopathology in the domain of interpersonal functioning. Scores range from 0 to 4. Lower scores mean a worse outcome.
Time Frame: 15 months
Population: These are the number of subjects for whom data was available for this measure during the relevant time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMI-PACT | Usual Care
Number analyzed (Participants) | 162 | 165
score on a scale | 2.42 (0.89) | 2.39 (0.89)

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Arm/Group | SMI-PACT | Usual Care
All-Cause Mortality (participants affected / at risk) | 3/164 | 1/167
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/167
Other Adverse Events (participants affected / at risk) | 0/164 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT01668355/Prot_SAP_000.pdf